CLINICAL TRIAL: NCT06741436
Title: Identification of Early HFpEF After Preeclampsia by Exercise Stress Testing
Brief Title: Exercise Testing After Preeclampsia
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Kathryn Lindley, Dr. Kathryn Lindley, MD, FACC, Vanderbilt University Medical Center
Other Study IDs: U13728
Record Dates: First submitted 2024-12-09; First posted 2024-12-19 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-01

CONDITIONS: Preeclampsia; Heart Failure Preserved Ejection Fraction; Hypertension
Keywords: CPET; Placental vascular dysfunction; echo
MeSH Terms: conditions — Pre-Eclampsia; Heart Failure, Diastolic; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of cord blood, placenta, urine, and venous blood will be collected and stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: Controls who meet the same inclusion/exclusion criteria, except they do not have preeclampsia and do not have pre-existing diabetes or chronic hypertension.
- PreE Px: Preeclamptic participants who meet the inclusion/exclusion criteria

SUMMARY:
Though cardiovascular disease (CVD) is the leading cause of mortality in women, traditional epidemiology in this area has focused on later life, when cardiometabolic risk has already exacted a cumulative toll on the vascular system. Recent data from the investigators and others has highlighted pregnancy as a unique, early moment of cardiovascular stress in young women that may "unmask" CVD propensity. It is unclear if PreE simply represents a "failed stress test" or directly contributes to the pathophysiology of future CVD. While mechanistic studies have largely been the purview of model-based studies, endothelial dysfunction has emerged as central to the pathogenesis of both PreE and peripartum cardiac dysfunction. Indeed, biomarkers of endothelial dysfunction and angiogenic imbalance during pregnancy have been shown to remain elevated at least 6 months post-partum. Moreover, peri-partum endothelial dysfunction can persist for years post-delivery and remains a significant risk factor for CVD (even after adjustment for other traditional risk factors). While these findings suggest that PreE-associated endothelial dysfunction and inflammation may contribute to early myocardial dysfunction that presages HF risk decades before its onset, the modifiable epidemiology of PreE-associated LVDD, including potential mechanisms of risk, remains unclear, limited by lack of precision molecular phenotypes accessible in a large number of American women across race. Ultimately, understanding the epidemiology and pathobiology of PreE-associated myocardial dysfunction affords a unique opportunity to identify women at risk with a longer lead-time for risk factor modification to interrupt CVD.

The investigators hypothesize that persistent structural-functional myocardial alterations after PreE are linked to pre- and post-gravid cardiometabolic risk factors (SA1), functional and hemodynamic impairment (SA2) and select pathways of vascular and inflammatory stress relevant to HF risk (SA3). Despite extensive study on the role of inflammation/ischemia in PreE, there have been no large studies connecting these phenotypes with early PP functional response and biochemical alterations, a key barrier to designing studies for improving CVD/HF in women.

SA1: To identify pregnancy-specific clinical factors related to postpartum HFpEF phenotypes Clinical Implication: Improve identification of women at highest risk for developing post-PreE LV diastolic dysfunction (a harbinger of HFpEF).

SA2: To define functional and hemodynamic signatures of early HFpEF due to preeclampsia

Clinical Implication: Identify women at highest risk for developing early HFpEF.

SA3: To identify shared pathophysiologic mechanistic pathways for PreE-associated HFpEF Clinical Implication: Identify targetable pathways for post-PreE cardiac dysfunction that may prevent/ delay HFpEF development.

DETAILED DESCRIPTION:
Participants will be identified by daily electronic health record (EHR) search with American College of Obstetricians and Gynecologists (ACOG) criteria for PreE. The investigators will begin recruitment of participants in both their third trimester, as well as at admission to the Labor and Delivery Service. The investigators may consent and enroll patients in the study prior to being admitted, to allow ample time to consider participation. Patients admitted to the Labor and Delivery service will be identified as being diagnosed with PreE using a checklist, with supervision of a board-certified obstetrician with NIH- funded experience in obstetric research.

Participants will be recruited and enrolled until the investigators reach the goal of 250 cases and 250 controls. The subject will first be prescreened for eligibility. The study team will then approach the care team of the subject and request permission to approach the subject about participation in the study. Once permission has been granted the study team will then approach the subject.

Once the study team is in contact with the potential participant (and it has been assessed that they meet study eligibility), they will receive a complete explanation of the protocol, and the informed consent will be reviewed with them. The consent form will clearly state that participants may end participation at any time without prejudice, and this is emphasized to the subject. In particular, participants who receive their health care at Vanderbilt University Medical Center will be reassured that their decision to decline participation will in no way affect their medical treatment.

In order to assess the capacity to consent in critically ill patients, a member of the study team will ask the participants about their understanding/awareness of their condition and their perceived reason for their hospitalization. If the study team suspect impaired competence based on subject's responses, the subject will be excluded from the study.

Enrollment. For this study, the investigators will leverage the multidisciplinary cardio-obstetrics clinical research team, a collaboration between the Cardiology Division, Dept of Medicine and Maternal Fetal Medicine, Dept of Obstetrics and Gynecology established and led by PI Lindley. The team is designed to deploy high-success methods to recruit, schedule, follow-up and retain participants. At Vanderbilt University Hospital, there are >5000 deliveries per year; of these, 22% women develop hypertensive disorders of pregnancy. The investigators have previously been very successful in recruiting patients with PreE from both the Women's Health Clinic, and the inpatient Labor and Delivery service, and anticipate no difficulties with recruitment. PI Lindley has previously successfully recruited over 350 postpartum women with hypertensive disorders of pregnancy for prospective clinical studies and has previously successfully completed a pilot study of postpartum exercise stress testing at 12-16 weeks after delivery in 53 women with PreE, with 49% racial/ethnic minority women recruited and retained. For this study, the goal is that ~25% of enrolled participants would self-identify as black.

Dr. Lindley is also the PI on the 'Multi-Omics for Maternal Health after Preeclampsia' (MOM-Health) study (IRB # 232160). In the event that participants choose to co-enroll in both studies, the investigators may use data from MOM-Health and vice versa to reduce duplication of study procedures where there may be overlap (ex: Biospecimen collection, surveys etc.). Study staff will strive to match up co-enrolled participants' follow-up visits so that they may be homogenized into one visit.

Surveys and questionnaires (At enrollment/ Within ~48 hr. of delivery, approximately 12-16 weeks postpartum, and approximately 1 year postpartum): The questionnaires regarding demographics, medical history, breastfeeding and reproductive health, substance use, mental health and functional status will be obtained.

Cardiovascular Assessment (within approximately 48 hr. of delivery, approximately 12-16 weeks postpartum, and approximately 1 year postpartum): Participants will have vital signs (blood pressure, heart rate, weight) obtained at each visit. In addition, either at enrollment during the third trimester, or prior to discharge from delivery hospitalization, participants will be given an at home blood pressure monitor with instructions on how to use the blood pressure cuff and report results. Participants will be asked to take their blood pressure up to twice per day, every day (morning and afternoon/evening), with instructions to retest within 15 minutes if an elevated blood pressure is detected. Blood pressure readings will be self-recorded, using an EHR log provided to the subject (My Health at Vanderbilt blood pressure flowsheet). Alternatively, participants will use a Bluetooth enabled device that allows the blood pressure readings to be directly transmitted into the EHR, viewable by their providers and study staff. Participants who forget to measure their blood pressures will be gently reminded to continue to do so. Participants will not be asked to return the cuff (it is theirs to keep). If they lose the cuff, the investigators will give them a replacement.

Brachial artery reactivity testing (BART) (approximately 12-16 weeks postpartum and approximately 1 year postpartum): the investigators will perform BART on all participants to assess PP endothelial function. Technique: Patients will be placed in the supine position with a blood pressure cuff in place on the upper arm. The brachial artery will be imaged with ultrasound. Baseline flow will be estimated by pulsed Doppler. Subsequently, the cuff will be inflated to 50 mmHg above systolic pressure, then released. Pulsed Doppler measurements of the brachial artery will be recorded every 30 seconds until 2 minutes after release of occlusion. Flow mediated dilatation (FMD) will be assessed by maximal percent change from baseline to post-inflation velocity. The investigators have experience in acquisition of these measures during exercise in the PP setting, increasing feasibility.

Rest echocardiography (within approximately 48 hr. of delivery, approximately 12-16 weeks postpartum, and approximately 1 year postpartum): Initial echocardiography will be obtained at the bedside on the Labor and Delivery unit at enrollment (within approximately 48 hours of delivery) and again at approximately 12-16 weeks postpartum, and approximately 1 year postpartum.

Perturbational echocardiography (approximately 12-16 weeks postpartum and approximately 1 year postpartum): In addition to rest echocardiography, the investigators will perform two sets of perturbations aimed at providing a volume challenge (leg lift) and assessing response to exercise (CPET). The investigators will be following ACC/AHA guidelines for performance/termination of exercise testing, and as such, these measures are safe in the postpartum setting.

* Leg lift: The protocol proposed here has been employed in large NHLBI studies to unmask early HFpEF predisposition in the Multi-Ethnic Study of Atherosclerosis (MESA) cohort. Passive leg raise will be performed for 2 minutes on a 45o wedge for a volume load. Passive leg raise maneuver does not carry any significant risk to the patient.
* Exercise (CPET): After leg lift echocardiography acquisition is complete, study participants will sit upright and allowed to recover for approximately 15 minutes. The investigators will next perform CPET with echocardiography at peak exercise. CPET will be performed on an upright cycle ergometer or treadmill per this protocol. Participants will be monitored by 12-lead electrocardiogram throughout exercise. Participants can choose to cease exercise before peak effort is reached, and individuals will be continuously monitored with "stopping rules" in place to limit risk of exercise-related complications (e.g., arrhythmia, HTN, hypotension), as noted by ACC/AHA guidelines on exercise testing. Echocardiography will be obtained in the upright position at peak exercise.

Biomarkers of placental vascular dysfunction and inflammatory stress (within approximately 48 hr. of delivery, approximately 12- 16 weeks postpartum, and approximately 1 year postpartum): Within approximately 48 hours of delivery, approximately 12- 16 weeks postpartum, and approximately1 year postpartum, the investigators will collect up to 50 ml of maternal venous blood which will be centrifuged and frozen at -80°C until use. As in the preliminary work, sFLT-1 and PIGF will be analyzed by ELISA. The investigators have also enlisted a less targeted approach to provide broader insight into inflammation, microvascular ischemia and endothelial dysfunction that characterize PreE-induced HFpEF, using the Olink system. The obtained placental, cord blood and urine samples obtained at delivery will be stored as resources in the cardiovascular biobank for future investigative studies by the scientific community to increase the impact of the investment of the participants. Urine samples will be obtained at each additional follow-up. Although no immediate genetic testing is planned for the specimens collected in this study, studies relating to genetic risk factors for cardiovascular disease/hypertensive disorders of pregnancy may perform genetic testing on these specimens in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Women age > 18 years
2. Give birth at VUMC
3. Have a diagnosis of PreE based on accepted American College of Obstetricians and Gynecologists criteria

Exclusion Criteria:

1. Age <18 years old
2. Unable to provide informed consent
3. Does not speak English
4. Active COVID-19 infection
5. Residual symptoms related to prior COVID-19 infection
6. HIV infection
7. Hepatitis B or C infection
8. Pulmonary arterial hypertension
9. Sickle cell disease
10. Pulmonary embolism
11. Pre-existing cardiomyopathy
12. Coronary artery disease
13. Active substance abuse (other than tobacco or marijuana)
14. Unable to attend postpartum visits

Controls

1. Enrolling controls who meet the same inclusion/exclusion criteria, except they do not have preeclampsia and do not have pre-existing diabetes or chronic hypertension.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population will include women who can biologically bear children. Traditionally, women (especially minorities) have been under-represented in studies to characterize HFpEF predisposition, despite their disproportionate risk. VUMC is located in the Southeast and cares for a disproportionate number of Black pregnant women with Preeclampsia. Given the increased risk of PreE in Black populations, we strive to maximize enrollment of Black women in our study, with a target of at least 25% of the enrolled subjects self-identifying as Black. Our targeted enrollment of Black women addresses clinical and investigative gaps in this population at high short and long-term CV risk following a preeclamptic pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
To measure relation between postpartum subclinical LV diastolic dysfunction and pregnancy-specific risk factors in 250 women with PreE and 250 normotensive women through echocardiographic imaging. | 12 months
  Pre-pregnancy risk factors (HTN, DM, delivery body mass index [BMI], age), pregnancy-specific risk factors (PreE severity, gestational age at delivery, gravidity, GDM, SGA) and PP risk factors (weight change, median systolic BP 0-2 weeks PP, resting BP at study visit) will be measured. Ordinary least squares (OLS) regressions will be used to estimate the relationship between Lateral E/e' at 52 weeks and the above risk factors, adjusting for baseline values, to determine if the diastolic function parameters are affected by the risk factors of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Lindley, MD, FACC, Principal Investigator — VUMC
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No